CLINICAL TRIAL: NCT06275087
Title: Differences in Speed of Recovery From Anesthesia and Recovery of Muscle Strength in General Balanced Inhalation Anesthesia and Total Intravenous Anesthesia for Intraoral Surgery - Clinical Randomised Trial
Brief Title: Differences in Speed of Recovery From Anesthesia for Intraoral Surgery
Acronym: PSIOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Ivan Šitum, MD, Principal invesigator, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: situm1phd
Record Dates: First submitted 2024-02-09; First posted 2024-02-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Intraoral Tumor
Keywords: TIVA; Propofol; Intraoral surgery; Postoperative recovery; recovery of muscle strenght
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA group (Experimental): The study involves patients in an operating room undergoing standard procedures. The induction procedure for anesthesia is the same for both groups, using sufentanil, propofol, and cisatracurium.
  In the TIVA group, anesthesia is maintained with continuous propofol infusion and intermittent cisatracurium doses, guided by neuromuscular and electroencephalogram monitoring. At the end of surgery, neuromuscular block is reversed, and extubation occurs when the train-of-four (TOF) index is over 90%.
  Muscle strength and bite force are measured at different intervals before and after anesthesia, using specific instruments. Additionally, patients fill out the Quality of recovery-40 (Qor-40) questionnaire at various time points to assess the quality of recovery after surgery and anesthesia.
  Interventions: Drug: Propofol
- Volatile group (Active Comparator): In the volatile group, anesthesia is maintained with inhaled sevoflurane and intermittent cisatracurium doses. Cisatracurium is repeated based on TOF ratio, and anesthesia depth is controlled by BIS, maintaining values between 25 and 50. Drug doses are adjusted according to TOF and BIS values.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — The experimental group will not receive volatile anesthetic, instead, they will receive propofol infusion
  Other Names: TIVA
  Arms: TIVA group
Drug: Sevoflurane — The control group will not receive TIVA, instead, they will receive sevoflurane via inhalation
  Other Names: general volatile anesthesia
  Arms: Volatile group

SUMMARY:
The goal of this clinical trial is to compare two groups of patients going in general anesthesia for intraoral surgery, the first group TIVA with propofol and the second group inhalational with sevoflurane. The main questions it aims to answer are to asses speed and quality of recovery from general anesthesia.

Participants will fill out a questionnaire to evaluate the quality of recovery from anesthesia using the QoR-40 1h, 24h, and 30 days after waking up from anesthesia in comparison to the results of the same questionnaire before surgery. Also, the investigators will perform a hand grip and bite strength test on the patients after waking up from anesthesia in the operating room, after 1 hour in the recovery room, and after 24 hours compared to preoperative values.

The investigators will compare TIVA and Volatile groups to see if there are any differences in recovery seed, muscle strength recovery, postoperative nausea and vomiting, and shivering between groups.

DETAILED DESCRIPTION:
After obtaining the approval of the ethics committee of KBC Zagreb and the Faculty of Dentistry of the University of Zagreb, the research will be conducted at KBC Zagreb.

Criteria for patient inclusion are:

* patients older than 18 years
* ASA status 1-2,
* Patients who have an indication for an intraoral surgical procedure (intraoral tumor excisions) longer than 30 minutes.
* patients who agreed to the research and signed the consent

Exclusion criteria are:

* ASA status 3 and higher,
* The need for postoperative care in the ICU,
* Surgery lasting more than 2 hours,
* Surgical procedures that in the operative plan include injuries to the grip of the masticatory muscles, the masticatory muscles themselves, and procedures on the bone, and thus may result in a difference in the strength of the bite. Masticatory muscles are defined as musculus pterygoideus lateralis, musculus pterygoideus medialis, musculus temporalis and musculus masseter.
* Surgical procedures on the bone where the bite force test alone could cause injury
* Patients with diseases of the neuromuscular junction and muscle diseases, myopathy, dystrophy
* Patients taking medications that can cause myopathy or muscle weakness
* Known allergies to drugs used in the trial,
* Refusing to participate

Participants will be randomly divided (1:1 randomisation) according to a predetermined randomization table (32) into the TIVA group and the Volatile group. After identification of the participants in the operating room, participants will be fitted with a peripheral venous line, electrocardiogram monitoring, non-invasive blood pressure measurement, pulse oximeter, capnograph, temperature probe, and bispectral index (BIS) of the electroencephalogram and neuromuscular monitoring, kinemiography with train-of-four (TOF , M-NMT, Drägerwerk AG & Co. KGaA,) by recording the responses.

The initial anesthesiological induction procedure will not differ in both groups of patients. The drugs that will be used are sufentanil 0.3mcg/kg, propofol 2mg/kg, and cisatracurium 0.1mg/kg.

Participants will be intubated with an endotracheal tube and mechanically ventilated with a mixture of oxygen and air (inspiratory fraction of oxygen 40%) with a total flow of gas mixture of 3 L/min.

Anesthesia will be maintained in the volatile group with the inhaled anesthetic sevoflurane and single doses of cisatracurium. Cisatracurium will be repeated when the TOF ratio is greater than 5%, and the repeat dose will be 0.01 mg/kg. The depth of anesthesia will be controlled by BIS, maintaining values between 25 and 50. Recommended drug doses will be guided by TOF and BIS values.

In the TIVA group, anesthesia will be maintained with a continuous infusion of propofol (5-10 mg/kg/h) and single doses of cisatracurium. Cisatracurium will be repeated when the TOF ratio is greater than 5%, and the repeat dose will be 0.01 mg/kg. The depth of anesthesia will be controlled by BIS, maintaining values between 25 and 50. Recommended drug doses will be guided by TOF and BIS values.

At the end of the surgical intervention in both groups, the neuromuscular block will be antagonized with prostigmine (0.05 mg/kg) along with atropine (0.01 mg/kg) as soon as the patient begins to breathe spontaneously. Patients will then be extubated when the TOF index is greater than 90%

Muscle strength of all participants will be measured with a JAMAR hand dynamometer, and bite force with a gnathodynamometer (Bite force sensor, Monad electronics) in four time intervals:

1. Before introduction to anesthesia
2. After waking up from anesthesia in the operating room
3. 1 hour after waking up from anesthesia in the recovery room
4. After 24 hours from the operation

All patients will fill out the Quality of recovery-40 (Qor-40) questionnaire for assessing the quality of recovery after anesthesia and surgery in four time intervals:

1. Before introduction to anesthesia
2. 1 hour after waking up from anesthesia in the recovery room
3. After 24 hours from the operation
4. After 30 days from the operation Consent for the use of the QoR-40 questionnaire was obtained by the main researcher from the author, Professor P.S. Myles, and Dr. M. Miklić Bublić, who translated the questionnaire into Croatian.

Postoperative nausea and vomiting and postoperative shivering will also be recorded, as a binary outcome (yes/no), by visual assessment and interaction with the patient.

The time from the end of the operation to waking up will be monitored. Pain will also be recorded based on QoR40 and the visual analogue scale (VAS-scale) for pain assessment. The patient's chronic therapy is recorded, as is the need for postoperative analgesia.

Assuming medium to large effect size, test power of 80% and use of independent t-test for the primary objective and x2 test for the secondary objective with a statistical significance of 0.05, it is necessary to take a sample of 42 patients, 21 subjects per group. . The test for power calculation is G Power Version 3.1.9.6 (46). Assuming that part of the respondents will not be able to follow up until the end of the research, a sample of 50 patients will be taken, that is, 25 patients in each group. A review of similar studies confirmed the sample size (18,47,48). The results will be processed with IBM SPSS statistics v27. For scalar parametric data, the independent Student t test will be used, for non-parametric data, the Mann-Whitney U test, while categorical data will be processed with the Pearson χ² test. One interim analysis for feasibility and precision estimation is planned.

ELIGIBILITY:
Criteria for patient inclusion are:

* patients older than 18 years
* ASA status 1-2,
* Patients who have an indication for an intraoral surgical procedure longer than 30 minutes.
* Surgical interventions on the soft tissues of the mouth, intraoral excision of tumors, operated through the transoral route
* Patients who agreed to the research and signed the consent

The exclusion criteria are:

* ASA status 3 and higher,
* The need for postoperative care in the ICU,
* Surgery lasting more than 2 hours,
* Surgical procedures that in the operative plan include injuries to the grip of the masticatory muscles, the masticatory muscles themselves, and procedures on the bone, and thus may result in a difference in the strength of the bite. Masticatory muscles are defined as musculus pterygoideus lateralis, musculus pterygoideus medialis, musculus temporalis and musculus masseter.
* Surgical procedures on the bone where the bite force test alone could cause injury
* Patients with diseases of the neuromuscular junction and muscle diseases, myopathy, dystrophy
* Patients taking medications that can cause myopathy or muscle weakness
* Known allergies to drugs used in the trial,
* Refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
"Quality of recovery from anesthesia" QoR-40 questionnaire | 1 hour, 24 hour, 30 day
  The QoR-40 is a recovery-specific and patient-rated questionnaire that contains 40 items measuring five dimensions: the physical comfort (12 items), emotional state (nine items), physical independence (five items), psychological support (seven items) and pain (seven items). The total score and subscales of the QoR-40 are measured using a five-point Likert scale (for positive items: 1 = none of the time, 5 = all of the time; for negative items, the scoring was reversed) and individual scores are then added together, with the minimum score being 40 points and the maximum score being 200 points. The QoR-40 was specifically designed to measure a patient's health status after surgery and anesthesia, and its completion time generally ranges from three to 10 min. The Japanese version of the QoR-40 was also validated according to standard methods of cultural adaptation and psychometric analysis in 2011.

SECONDARY OUTCOMES:
bite strength and hand grip strength | after waking in OR up to 10 min, 1 hour after waking, 24 hour after waking
  Hand-grip muscle strength and bite strength will be measured with a dynamometer on three occasions: before general anesthesia, in the early post-anesthesia period in the operating room, and 24 hours after anesthesia.
Postoperative nausea and vomiting | 24 hours
  determine the difference in the frequency of postoperative nausea and vomiting
Postoperative shivering | 2 hour
  determine the difference in the frequency of postoperative shivering

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Šitum, MD, Principal Investigator — UHC Zagreb
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
If there is a need and desire on the part of other researchers, data on patients without personal data can be shared

REFERENCES:
- [Background] Diniz JA, Siqueira ADS, Araujo GM, Faro TF, Torres LHS, Oliveira E Silva ED, Laureano Filho JR. Intraoral Approach for Surgical Treatment of Psammomatoid Juvenile Ossifying Fibroma. J Craniofac Surg. 2020 May/Jun;31(3):e306-e309. doi: 10.1097/SCS.0000000000006171. PMID 31934971
- [Background] Ferreira, C. C., Pereira, M. B. F., Bruzinga, F. F. B., Castro, H. H. O., Souto, G. R., Souza, P. E. A., & De Oliveira, L. J. (2022, September). AN UNUSUAL INTRAORAL LIPOMA: A CASE REPORT. Oral Surgery, Oral Medicine, Oral Pathology and Oral Radiology, 134(3), e119. https://doi.org/10.1016/j.oooo.2022.01.212
- [Background] Frerich, B. (2020). Complications in Maxillofacial Tumor Surgery. Complications in Cranio-Maxillofacial and Oral Surgery, 253-277. https://doi.org/10.1007/978-3-030-40150-4_13
- [Background] Tamunobelema, D. M. S., & Uruaka, C. I. (2023, March 11). General Anaesthetic Agents and its Implication on the Cardiovascular System: A Systemic Review. Saudi Journal of Medical and Pharmaceutical Sciences, 9(03), 171-183. https://doi.org/10.36348/sjmps.2023.v09i03.006
- [Background] Qurbani, B., & Karim, S. B. (2022, December 29). Comparison among complications of common intravenous anesthetic drugs during general anesthesia for patients undergoing surgery in Sulaimani city. Annals of the College of Medicine, Mosul, 44(2), 159-165. https://doi.org/10.33899/mmed.2022.136178.1166
- [Background] Fiorda-Diaz, J., Stoicea, N., & Bergese, S. (2017). Anesthetic Agents. Essentials of Neuroanesthesia, 123-129. https://doi.org/10.1016/b978-0-12-805299-0.00007-5
- [Background] Hao X, Ou M, Zhang D, Zhao W, Yang Y, Liu J, Yang H, Zhu T, Li Y, Zhou C. The Effects of General Anesthetics on Synaptic Transmission. Curr Neuropharmacol. 2020;18(10):936-965. doi: 10.2174/1570159X18666200227125854. PMID 32106800
- [Background] Monisha, B., Madhusudhana, R., & Sujatha, M. (2023). Effects of Isoflurane versus Propofol for Postoperative Neurocognitive Recovery in Patients Undergoing Surgery under General Anaesthesia: A Randomised Clinical Study. JOURNAL OF CLINICAL AND DIAGNOSTIC RESEARCH. https://doi.org/10.7860/jcdr/2023/62147.17888
- [Background] Mayhew D, Mendonca V, Murthy BVS. A review of ASA physical status - historical perspectives and modern developments. Anaesthesia. 2019 Mar;74(3):373-379. doi: 10.1111/anae.14569. Epub 2019 Jan 15. PMID 30648259
- [Background] Saha, D. S. C., & Seraji, D. S. I. (2023, April 16). A Comparative Study of Propofol and Sevoflurane for General Anesthesia in Laparoscopic Appendectomy. Scholars Journal of Applied Medical Sciences, 11(04), 753-757. https://doi.org/10.36347/sjams.2023.v11i04.014
- [Background] Yang L, Chen Z, Xiang D. Effects of intravenous anesthesia with sevoflurane combined with propofol on intraoperative hemodynamics, postoperative stress disorder and cognitive function in elderly patients undergoing laparoscopic surgery. Pak J Med Sci. 2022 Sep-Oct;38(7):1938-1944. doi: 10.12669/pjms.38.7.5763. PMID 36246684
- [Background] Miao L, Lv X, Huang C, Li P, Sun Y, Jiang H. Long-term oncological outcomes after oral cancer surgery using propofol-based total intravenous anesthesia versus sevoflurane-based inhalation anesthesia: A retrospective cohort study. PLoS One. 2022 May 13;17(5):e0268473. doi: 10.1371/journal.pone.0268473. eCollection 2022. PMID 35559987
- [Background] Zhou, Y., & Xu, T. (2022, January 24). Effect of propofol and sevoflurane on perioperative and postoperative outcomes in lung cancer patients after thoracoscopic surgery. Tropical Journal of Pharmaceutical Research, 20(4), 873-879. https://doi.org/10.4314/tjpr.v20i4.30
- [Background] Wu L, Li Y, Si J. Effects of sevoflurane and propofol on postoperative nausea and vomiting in patients with colorectal cancer placed under general anesthesia: a systematic review and meta-analysis. J Gastrointest Oncol. 2022 Dec;13(6):2963-2972. doi: 10.21037/jgo-22-783. PMID 36636047
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Miklic Bublic M, Miklic P, Barl P, Matas M, Sekulic A. CROATIAN VERSION OF THE QUALITY OF RECOVERY QUESTIONNAIRE (QoR-40): TRANSCULTURAL ADAPTATION AND VALIDATION. Acta Clin Croat. 2021 Jun;60(2):237-245. doi: 10.20471/acc.2021.60.02.09. PMID 34744273
- [Background] Kim DH, Min KT, Kim EH, Choi YS, Choi SH. Comparison of the effects of inhalational and total intravenous anesthesia on quality of recovery in patients undergoing endoscopic transsphenoidal pituitary surgery: a randomized controlled trial. Int J Med Sci. 2022 Jun 13;19(6):1056-1064. doi: 10.7150/ijms.72758. eCollection 2022. PMID 35813289
- [Background] Meng W, Yang C, Wei X, Wang S, Kang F, Huang X, Li J. Type of anesthesia and quality of recovery in male patients undergoing lumbar surgery: a randomized trial comparing propofol-remifentanil total i.v. anesthesia with sevoflurane anesthesia. BMC Anesthesiol. 2021 Dec 1;21(1):300. doi: 10.1186/s12871-021-01519-y. PMID 34852781
- [Background] Shi CM, Zhou Y, Yang N, Li ZQ, Tao YF, Deng Y, Guo XY. [Quality of psychomotility recovery after propofol sedation for painless gastroscopy and colonoscopy]. Beijing Da Xue Xue Bao Yi Xue Ban. 2023 Apr 18;55(2):324-327. doi: 10.19723/j.issn.1671-167X.2023.02.017. Chinese. PMID 37042144
- [Background] Kim SH, Ju HM, Choi CH, Park HR, Shin S. Inhalational versus intravenous maintenance of anesthesia for quality of recovery in patients undergoing corrective lower limb osteotomy: A randomized controlled trial. PLoS One. 2021 Feb 19;16(2):e0247089. doi: 10.1371/journal.pone.0247089. eCollection 2021. PMID 33606764
- [Background] Tomita S, Matsuura N, Ichinohe T. The combined effects of midazolam and propofol sedation on muscle power. Anaesthesia. 2013 May;68(5):478-83. doi: 10.1111/anae.12172. Epub 2013 Mar 22. PMID 23521655
- [Background] Wen LL, Lin WQ, Zhao WX, Li GC, Bai XH, Xiao JB. [Effect of sevoflurane versus propofol-remifentanil anesthesia on neuromuscular blockade by continuous cisatracurium infusion]. Nan Fang Yi Ke Da Xue Xue Bao. 2010 Jan;30(1):163-5. Chinese. PMID 20118012
- [Background] Man, Mi, & Han. (2011, September 1). Influence of sevoflurane and propofol on the neuromuscular block effect of cisatracurium. Medical Journal of Chinese People's Liberation Army, 36, 973-975. https://www.semanticscholar.org/paper/Influence-of-sevoflurane-and-propofol-on-the-block-Man-Mi/eb40663a5683c9cc22116520104ca02a66c8b6de#citing-papers
- [Background] Pan, C., Xing, Y., Zhang, D., Liu, X., Zhou, Y., Shi, L., Xu, M., & Zhang, B. (2023, June 6). Combined remifentanil/sevoflurane in paediatric tonsil surgery anesthesia: Effect on recovery time of respiration and consciousness in paediatric patients. Tropical Journal of Pharmaceutical Research, 22(5), 1073-1079. https://doi.org/10.4314/tjpr.v22i5.20
- [Background] Interlandi C, Di Pietro S, Costa GL, Spadola F, Iannelli NM, Macri D, Ferrantelli V, Macri F. Effects of Cisatracurium in Sevoflurane and Propofol Requirements in Dog-Undergoing-Mastectomy Surgery. Animals (Basel). 2022 Nov 14;12(22):3134. doi: 10.3390/ani12223134. PMID 36428361
- [Background] Liu J, Yang L. Effects of propofol and sevoflurane on blood glucose, hemodynamics, and inflammatory factors of patients with type 2 diabetes mellitus and gastric cancer. Oncol Lett. 2020 Feb;19(2):1187-1194. doi: 10.3892/ol.2019.11201. Epub 2019 Dec 10. PMID 31966048
- [Background] ALKAYA SOLMAZ, F., & KIRDEMİR, P. (2020, March 2). Enhanced recovery after surgery (ERAS) and anesthesia. Acta Medica Alanya, 4(1), 95-101. https://doi.org/10.30565/medalanya.587027
- [Background] Bennett J, McDonald T, Lieblich S, Piecuch J. Perioperative rehydration in ambulatory anesthesia for dentoalveolar surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Sep;88(3):279-84. doi: 10.1016/s1079-2104(99)70028-4. PMID 10503854
- [Background] Pollard BJ, Bryan A, Bennett D, Faragher EB, Un EN, Keegan M, Wilson A, Burkill M, Beatty PC, Stollery BT, et al. Recovery after oral surgery with halothane, enflurane, isoflurane or propofol anaesthesia. Br J Anaesth. 1994 May;72(5):559-66. doi: 10.1093/bja/72.5.559. PMID 8198909
- [Background] Asakura A, Mihara T, Goto T. The Effect of Preoperative Oral Carbohydrate or Oral Rehydration Solution on Postoperative Quality of Recovery: A Randomized, Controlled Clinical Trial. PLoS One. 2015 Aug 28;10(8):e0133309. doi: 10.1371/journal.pone.0133309. eCollection 2015. PMID 26317629
- [Background] Pocock SJ. Clinical Trials: A Practical Approach. Wiley; in 1983
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823